CLINICAL TRIAL: NCT05744778
Title: The Effect of Dry Needling Treatment Combined With Physical Therapy in Patients With Cervical Spondylosis: A Randomized Controlled Study
Brief Title: The Effect of Dry Needling Treatment Combined With Physical Therapy in Patients With Cervical Spondylosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Alper mengi, Medical Doctor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27.01.2023/15
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Dry Needling; Cervical Spondylosis; Physical Therapy
MeSH Terms: conditions — Spondylosis | interventions — Dry Needling; Physical Therapy Modalities; Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical therapy and rehabilitation (Experimental): The patient group who underwent physical therapy and rehabilitation.
  Interventions: Other: Physical therapy and rehabilitation
- Dry needling (Experimental): The patient group who underwent dry needling for trigger points in the upper trapezius muscle along with physical therapy and rehabilitation.
  Interventions: Other: Dry needling; Other: Physical therapy and rehabilitation

INTERVENTIONS:
Other: Dry needling — In addition to the physical therapy and exercise program, the dry needling group will consist of patients who have had 3 sessions of dry needling applied to the trigger points in the trapezius muscle, 5 days apart.
  Arms: Dry needling
Other: Physical therapy and rehabilitation — The physical therapy and rehabilitation group will consist of patients who will be applied the same exercise program together with the same physical therapy applications (superficial heat (infrared lamp), transcutaneous electrical nerve stimulation (TENS) and therapeutic ultrasound (TUS)) 5 sessions per week for 3 weeks.

SUMMARY:
In this study, it was aimed to determine whether dry needling treatment applied to the trigger points in the trapezius muscle in patients with chronic neck pain due to cervical spondylosis makes an additional contribution to the treatment results of the physical therapy and rehabilitation program.

DETAILED DESCRIPTION:
Among the evaluated patients, the patients meeting the inclusion and exclusion criteria will be randomized into 2 groups using the random numbers table.

While physical therapy and rehabilitation program will be applied to one group, dry needling treatment will be applied to the trigger points in the upper trapezius region with the same program to the other group. Patients will be evaluated before treatment (day 0) and at the end of treatment (day 21).

The randomization and evaluation of the patients will be done by Gül Tuğba Bulut, while the injection of the patients will be done by Alper Mengi.

Gender, age, education level, occupation, neck pain duration, body mass index of the patients included in the study will be recorded.

The patients will be evaluated in terms of pain intensity, number of active trigger points in the upper trapezius muscle, functional status, quality of life, anxiety and depression at before (day 0) and after treatment (day 21).

ELIGIBILITY:
Inclusion Criteria:

* Having neck pain for at least 3 months
* Restriction of neck movements and/or pain during movement
* Tenderness in neck paravertebral muscles and neural foramen with compression
* Detection of narrowing of intervertebral disc spaces, subchondral sclerosis, osteophyte on cervical radiograph
* Active trigger point in the upper trapezius muscle during the examination.

Exclusion Criteria:

* Having motor, sensory or reflex abnormalities due to spinal root compression
* Whiplash injuries
* Cervical spinal stenosis
* Having undergone cervical vertebra surgery
* History of interventional procedure on the cervical region in the last 6 months
* Central or peripheral nervous system disorders
* Spondylolisthesis
* Inflammatory neck pain
* History of infectious, chronic inflammatory disease, malignancy
* Not being cooperative
* Having open wounds, infections or sensory defects on the skin where the application will be made
* Fibromyalgia
* Advanced osteoporosis or osteomalacia
* Active psychiatric illness.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Pain severity | 1 day
  Pain intensity will be questioned by visual analog scale (VAS) as pain intensity at movement, rest, and night. A horizontal straight line 10 cm long will be used in the VAS assessment. 0 will be considered as no pain, 10 will be considered as the most severe pain. Movement pain will be questioned as the average of the pain felt while the patients are doing their daily routine, rest pain will be the average of the pain felt when the patients are not doing any activity during the day, and night pain will be the average of the neck pain when they wake up or wake up from sleep.

SECONDARY OUTCOMES:
Number of active trigger points | 1 day
  The upper trapezius muscle of the patient lying in the prone position will be examined and the location and number of active trigger points determined as a result of the examination will be recorded.
Functional status | 1 day
  The Neck Pain and Disability Scale (NPAD) will be used to measure the functional status of patients due to neck pain. NPAD consists of 20 questions including the effect of neck pain on emotional state and cognitive function and the relationship of neck pain with daily living activities. Each question takes a value between 0 and 5. Accordingly, 0 represents normal function and 5 represents the worst condition resulting from the pain problem. The total score of the scale, which takes a value between 0 and 100, is obtained by summing the scores of all questions.
Life quality | 1 day
  Short Form-12 (SF-12) will be used to evaluate the quality of life of the patients. SF-12 was created as a shorter form by taking 12 different items from 8 different subheadings of SF-36. It has 2 sub-parameters as physical and mental health. Higher scores indicate better health.
Anxiety and depression | 1 day
  Patients will be evaluated with the Hospital Anxiety and Depression Score (HADS) in terms of anxiety and depression. HADS consists of 14 questions in total. The minimum score for the anxiety and depression subscales is 0, and the maximum score is 21. An increase in the score on the scale means that the severity of anxiety and depression increases. The cut-off points were determined as 10 for the anxiety subscale and 7 for the depression subscale.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No